CLINICAL TRIAL: NCT01895465
Title: Improvement in Urine Collection Methods in Children
Acronym: 0244-12-RMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, waisman yehezkel, Associate Professor, MD, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SCHNEIDER/7329
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Urinary Tract Infection; Unspecified Fever
Keywords: urine collection, contamination
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A slitted diaper (Experimental): An ordinary pediatric urine collection bag used in the ED that will be used together with the slitted diaper
  Interventions: Device: Slitted diaper

INTERVENTIONS:
Device: Slitted diaper — A diaper where a slit is made through which a urine collection bag is pulled through
  Other Names: Huggies, Pampers, etc.

SUMMARY:
The population of children presenting to the Emergency Department (ED) for treatment increases day by day, creating a further burden on the limited nursing staff and where many children and their parents are forced to wait many hours until their medical investigation ends. Part of the many hours waited are for various tests the patient has to undergo, where the urine test is one of the main ones.

Urinary tract infections in children are a common cause of death due to acute and chronic complications alike. Our study aims to test a urine collection method to see whether it reduces parents' and/or nursing staff's involvement and thereby reducing the urine sample's percentage of contamination.

DETAILED DESCRIPTION:
The study intends to explore whether on obtaining a pediatric urine sample by using a diaper in an innovative way can shorten the waiting time parents have to endure until an urine sample is perceived, and accordingly, the percentage of contamination in the samples obtained. The innovativeness introduced is that by using an ordinary everyday diaper, which is found in all marketing outlets, and by making a slit in the diaper where the pediatric urine collecting bag can be pulled out and thus allowing parents/care takers to see straight away whether urine has been given and thus cut back on opening and reopening of the diaper.

ELIGIBILITY:
Inclusion Criteria:

1. Children incapable of giving urine voluntarily in the Emergency Department
2. Children requiring an urine test
3. Children whose parents have agreed to take part in the research and have signed a consent form

Exclusion Criteria:

1. Children who have an immediate medical condition which requires catheterization
2. Parents who have declined taking part in the research
3. Children who give urine voluntarily
4. Children who do not need an urine test for their continued treatment

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Recording of time elapsed between physician's request for an urine test to be taken until obtained | 12 months

SECONDARY OUTCOMES:
Percentage of contamination in urine cultures obtained | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel